CLINICAL TRIAL: NCT03655210
Title: 4week, a Multicenter, Randomized, Double-blinded, Parallel, Therapeutic Confirmatory Clinical Trial to Evaluate the Efficacy and Safety of HL151 Versus Placebo in Perennial Allergic Rhinitis Patients
Brief Title: To Evaluate the Efficacy and Safety of HL151 Versus Placebo in Perennial Allergic Rhinitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_HL151_301
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): HL151(1Tab,Bepostatine salicylate) once a day, 4 weeks of treatment
  Interventions: Drug: HL151
- Placebo Comparator (Placebo Comparator): HL151 Placebo (1Tab,Placebo of Bepostatine salicylate) once a day, 4 weeks of treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HL151 — HL151(1Tab) once a day for 4 weeks of treatments
  Arms: Experimental
Drug: placebo — HL151 placebo(1Tab, Placebo of Bepostatine salicylate) once a day for 4 weeks of treatments
  Arms: Placebo Comparator

SUMMARY:
4week, a Multicenter, Randomized, Double-blinded, Parallel, Therapeutic confirmatory Clinical Trial

DETAILED DESCRIPTION:
4week, a Multicenter, Randomized, Double-blinded, Parallel, Therapeutic confirmatory Clinical Trial to Evaluate the Efficacy and Safety of HL151 versus Placebo in perennial allergic rhinitis patients

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, 19 years ≤ age
2. At least two years history of allergic rhinitis prior to participate in clinical trial
3. Patients with positive reaction for perennial allergen in tests(prick test or Intradermal test or MAST(Multiple Allergen Simultaneous Test) or Immuno CAP test) within 12 months
4. In visit 2, patients with over mean 5 points of the total reflective TNSS score per day (during the run-in period) (highest value 12 points)
5. Patients who can ability to record subject diary
6. Patients who agreed to maintain the same environment throughout the entire clinical trial period.
7. Written consent voluntarily to participate in this clinical trial after understanding and detailed explanation about this clinical trial

Exclusion Criteria:

1. Patients with non-allergic rhinitis
2. Patients with asthma due to the following diseases(but patients with mild and intermittent asthma are available to participate in clinical trials)

   * Within four weeks from the date of screening, patients who visit the emergency room or have been hospitalized within 12 weeks or
   * patients with asthma who need other treatment except short-acting Beta-efficient respiratory relaxants Inhalation
3. Patients with obstructive nasal polyp or severe deviated nasal septum
4. Patients who Within 12 weeks from the date of screening, had damage or surgery around nasal cavity
5. Patients with anamnesis in acute /chronic sinusitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Changes in total rTNSS(Reflective TNSS) score | Visit 2 (0 week), Visit 3 (2 weeks), Visit 4 (4 weeks)
  Changes in total rTNSS(Reflective TNSS) score at 4 weeks after clinical drug administration compared to baseline

SECONDARY OUTCOMES:
Changes in rTNSS(Reflective TNSS) score | Visit 2 (0 week), Visit 3 (2 weeks)
  Changes in rTNSS(Reflective TNSS) score at 2 weeks after clinical drug administration compared to baseline
Changes in iTNSS(Instananeous TNSS) score | Visit 2 (0 week), Visit 3 (2 weeks), Visit 4 (4 weeks)
  Changes in iTNSS(Instananeous TNSS) score at 2 weeks and 4 weeks after clinical drug administration compared to baseline
Changes in rTNSS(Reflective TNSS) score (Information recorded in the TNSS section of the diary included-Runny Nose,Sneezing,Itchy) | Visit 2 (0 week), Visit 3 (2 weeks), Visit 4 (4 weeks)
  Changes in rTNSS(Reflective TNSS) score (Information recorded in the TNSS section of the diary included-Runny Nose,Sneezing,Itchy) at 2 weeks and 4 weeks after clinical drug administration compared to baseline
Changes in iTNSS(Instananeous TNSS) score (Information recorded in the TNSS section of the diary included-Runny Nose,Sneezing,Itchy) | Visit 2 (0 week), Visit 3 (2 weeks), Visit 4 (4 weeks)
  Changes in iTNSS(Instananeous TNSS) score (Information recorded in the TNSS section of the diary included-Runny Nose,Sneezing,Itchy) at 2 weeks and 4 weeks after clinical drug administration compared to baseline
Investigator's assessment of overall treatment | Visit 4 (4 weeks)
  Investigator's assessment of overall treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided